CLINICAL TRIAL: NCT00727545
Title: Effect of Weekly Rice Fortification With Iron on Frequency of Anemia and Hemoglobin Concentration Among Children Attending Public Day Care Centers From Rio de Janeiro
Brief Title: Effect of Rice Fortification With Iron on Anemia Among Children
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Responsible Party: Ursula Viana Bagni, Universidade Federal do Rio de Janeiro
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UFRJ-1
Record Dates: First submitted 2008-07-30; First posted 2008-08-04 (Estimated); Last update posted 2008-08-06 (Estimated); Status verified 2008-07

CONDITIONS: Iron Deficiency Anemia
MeSH Terms: conditions — Anemia, Iron-Deficiency

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Other: iron bisglycine chelate; Other: placebo

INTERVENTIONS:
Other: iron bisglycine chelate
Other: placebo

SUMMARY:
This was a double-blind community-based trial, placebo controlled. During 16 weeks, children in the intervention group (GI, n=180) received iron fortified rice, and children in the control group (GC, n=174) received rice with placebo. Anemia was considered present when hemoglobin < 11.0g/dL. Comparison of mean variation on hemoglobin between groups was accessed by using Student's t-test. Hemoglobin concentration improved in both groups, with mean increase of 0.42 g/dL in GI (11.28±1.23 g/dL to 11.75±1.16 g/dL, p < 0.001), and 0.49 g/dL in GC (11.06±1.13 g/dL to 11.51±1.16 g/dL, p < 0.001). Anemia decreased (p < 0.01) in both groups (37.8% to 23.3% in GI and 45.4% to 33.3% in GC), with no differences between them. Hemoglobin increase was significantly higher in children who received total amount of iron ≥ 53.76 mg from fortified rice, compared to those who received less than this cut-off value (0.94 g/dl vs 0.39 g/dl p=0.03). The results suggest that this type of intervention can be useful in anemia control if fortified food intake is adequate.

ELIGIBILITY:
Inclusion Criteria:

* pre-school children attending public day care centers

Exclusion Criteria:

* sickle cell anemia, purpura

Ages: 12 Months to 60 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 385 (Actual)
Dates: Start 2006-03; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Hemoglobin in crease

CONTACTS AND LOCATIONS:
Locations (1):
- Public day care centers, Rio de Janeiro, Brazil